CLINICAL TRIAL: NCT04044378
Title: Famitinib Malate (SHR1020) Plus Camrelizumab (SHR 1210) Versus Famitinib Malate Alone Versus Famitinib Malate Plus Ifosfamide Locally Advanced, Unresectable or Metastatic Osteosarcoma Progression Upon Chemotherapy: A Phase Ib/II Randomized and Controlled Dose-Escalation Trial
Brief Title: Famitinib Plus Camrelizumab & Famitinib Alone & Famitinib Plus Ifosfamide in Advanced Osteosarcoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: toxicity
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 08; CSSG (Other: Chinese Sarcoma Study Group)
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Effect of Drugs; Progression; Pediatric Cancer
Keywords: famitinib; camrelizumab; advanced osteosarcoma; recommended phase 2 dose; efficacy; ifosfamide
MeSH Terms: conditions — Disease Progression; Neoplasms | interventions — famitinib; Ifosfamide; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: famitinib and camrelizumab (Experimental): In the dose-defining phase I portion, camrelizumab was given at a fixed dose of 200mg Q2W, while the de-escalated 3+3 design was used to detect the recommended dose of famitinib from an initial level of 15mg orally taken daily. Recommended phase 2 dose (RP2D) was defined as the highest dose at which no more than 30% patients experience a DLT in the first two courses.
  In the phase II portion, famitinib will be orally taken daily with RP2D together with camrelizumab intravenous infusion at a dose of 200 mg over 30 minutes, once every two weeks (Q2W), 4 weeks (28 days) as one treatment cycle.
  Interventions: Drug: Famitinib; Drug: Camrelizumab
- Arm B: famitinib alone (Active Comparator): Only phase II portion (Phase I have been completed): famitinib will be 20mg orally taken daily, 4 weeks (28 days) as one treatment cycle.
  Interventions: Drug: Famitinib
- Arm C: Famitinib and Ifofamide (Experimental): Only phase II protion (Phase I have been completed): famitinib will be 20mg orally taken daily, 4 weeks (28 days) as one treatment cycle together with ifofamide 1800 mg/m^2/day intravenous infusion will be administered on Days 1 to 3 and 15-17 of each 28-day cycle for a total of 5 cycles.
  Interventions: Drug: Famitinib; Drug: Ifosfamide

INTERVENTIONS:
Drug: Famitinib — famitinib with RP2D orally daily
Drug: Ifosfamide — ifosfamide 1.8g/m2/d d1-3, 15-17 Q4W infusion
  Arms: Arm C: Famitinib and Ifofamide
Drug: Camrelizumab — camrelizumab 200mg infusion once Q2W
  Other Names: camralizumab
  Arms: Arm A: famitinib and camrelizumab

SUMMARY:
Results of previous study showed high objective response but short-term activity of anti-angiogenesis tyrosine kinase inhibitors in advanced osteosarcoma. Given the recent success of immunotherapies, combinations of antiangiogenics with immune checkpoint blockers have become an attractive strategy. The investigators had completed an prospective phase 2 trial of the combination of apatinib and camrelizumab on advanced osteosarcoma and showed prolonged progression-free survival for this combination. Famitinib is a novel tyrosine kinase inhibitor targeting VEGFR-2, -3 and FGFR-1, -2, -3, -4 with high affinity, which showed broad antitumor activity against a variety of xenograft models.

A Study to Compare the Efficacy and Safety of Levatinib with or without Ifosfamide and Etoposide in Children, Adolescents and Young Adults With Relapsed and Refractory Osteosarcoma showed promising median PFS of 11.3 months. Thus we also try to investigate the combination efficacy of TKIs with chemotherapy in advanced osteosarcoma.

This study aims to investigate the recommended phase 2 dose for pediatric use of famitinib in combination with camrelizumab and trys to explore the efficacy and safety for single drug famitinib, famitinib and camrelizumab and famitinib and ifosfamide in patients with inoperable high-grade osteosarcoma progressing after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent and sign the informed consent form;
* ≥12 years old, male and female (For phase I portion, only 12-17 years old with 12 and 17 years old included; for phase II portion, more than 12 years old);
* Histopathologically or cytologically confirmed Advanced Osteosarcoma; (Local tumors and solitary pulmonary lesions must be confirmed by pathological diagnosis. Multiple pulmonary metastases need no pathological examination.)
* Failed to receive chemotherapy for osteosarcoma (including HD-MTX, anthracyclines, DDP and IFO) are defined as those who progress within 6 months after adjuvant chemotherapy and chemotherapy for advanced osteosarcoma, and those who progress over 6 months require the consent of the subject or his legal representative.;
* Have at least one measurable lesion (in accordance with RECIST v1.1, major diameter ≥10 mm of the measurable lesion in spiral CT scan or short diameter of swollen lymph node ≥15 mm; the lesion with previous local therapy can be used as target lesion after the progression is confirmed in accordance with RECIST v1.1);
* For subjects with progression after local regional therapy, the local regional therapy (including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic arterial infusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) must has been completed at least 4 weeks prior to baseline radiological scanning, and any toxicity (except alopecia) induced by local regional therapy must have resolved to ≤ Grade 1 in accordance with national cancer institute - common terminology criteria for adverse event version 4.03 (NCI-CTCAE v4.03);
* ECOG-PS score 0-1;
* With a life expectancy of ≥12 weeks;
* The body surface area is over 1.2 m2;
* Have the required screening laboratory values including the following parameters (within 7 days prior to the start of study treatment):
* Hematology: (except for hemoglobin, no blood transfusion or use of granulocyte colony-stimulating factor [G-CSF] or use of drugs for correction within 14 days prior to screening); Absolute neutrophil count ≥0.75×109/L; Platelet count ≥75×109/L; Hemoglobin ≥80 g/L;

Blood biochemistry: (no infusion of albumin within 14 days):

Serum albumin ≥25 g/L； Serum total bilirubin ≤1×upper limit of normal (ULN); Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (AKP) ≤2.5×ULN; Serum creatinine (Cr) ≤1.5×ULN or Cr clearance >50 mL/min (Cockcroft-Gault formula as below) Man: Cr clearance =((140-age) ×weight)/(72×serum Cr) Woman: Cr clearance =((140-age) ×weight)/ (72×serum Cr) × 0.85 Weight unit: kg; serum Cr unit: mg/mL;

* Women of childbearing potential: must agree on abstinence (avoid heterosexual intercourse) or use of contraception methods with annual contraceptive failure rate of < 1% following the signature of informed consent form until at least 120 days after the last dose of study drug. The serum human chorionic gonadotropin (HCG) test must be negative within 7 days prior to enrollment in the study; and the subjects must not be in lactating period.

If the female subject has menses, has not reached postmenopausal state (absence of menses for ≥ consecutive 12 months, with no other reason found except menopause) and has not received sterilization operation (e.g., hysterectomy, bilateral tubal ligation or bilateral ovariectomy), she would be considered to have childbearing potential.

Exclusion Criteria:

* Other active malignant tumor except advanced osteosarcoma within 5 years or simultaneously. Cured localized tumor, for example, basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate, carcinoma in situs of cervix, breast cancer in situ may be enrolled;
* History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage, for example, esophageal and fundal varices with hemorrhagic risk, locally active peptic ulcer, persistent fecal occult blood (+) (the fecal occult blood test can be repeated if it is positive at baseline, and gastroduodenoscopy [EGD] would be needed if it is still positive in repeated test; the patient can not be enrolled if the EGD shows esophageal and fundal varices with hemorrhagic risk);
* Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment;
* Known genetic or acquired hemorrhage (e.g., coagulation dysfunction) or thrombotic tendency, for example, patient with hemophilia; current or recent (within 10 days prior to the start of study treatment) use of full-dose of oral or intravenous anticoagulant or thrombolytic drug for the purpose of treatment (preventive use of low-dose aspirin or low molecular weight heparin is allowed);
* Current or recent (within 10 days prior to the start of study treatment) use of aspirin (> 325 mg/day) or dipyridamole, ticlopidine, clopidogrel and cilostazol;
* Thrombosis or thromboembolic event within 6 months prior to the start of study treatment, for example, cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism;
* Cardiac clinical symptom or disease that is not well controlled, for example, (1) > Grade II cardiac insufficiency in accordance with New York Heart Association (NYHA) criteria or color Doppler echocardiography: LVEF (left ventricular ejection fraction) <50%; (2) unstable angina pectoris; (3) myocardial infarction within one year prior to the start of study treatment; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) QTc > 450 ms (males) or QTc > 470ms (females) (QTc interval is calculated by Fridericia formula; In case QTc is abnormal, it can be detected for three times at an interval of 2 minutes and the average will be taken);
* Hypertension that can not be well controlled through antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) (based on the average of BP readings acquired from ≥2 measurements), allowing to reach the above parameters by the use of antihypertensive therapy; previous hypertensive crisis or hypertensive encephalopathy;
* Major vascular disease within 6 months prior to the start of study treatment (for example, aortic aneurysm requiring surgical repair or peripheral arterial thrombosis in recent days);
* Serious, uncured or splitting wound and active ulcer or untreated bone fracture;
* Major surgical therapy within 4 weeks prior to the start of study treatment (except diagnosis), or expected major surgery during the study;
* Inability or unwilling to swallow tablets, malabsorption syndrome or any condition affecting gastrointestinal absorption;
* Intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months prior to the start of study treatment, including incomplete obstruction that is related with the original disease or needs routine parenteral hydration, parenteral nutrition or tube feeding; If the subject has signs/symptoms of incomplete obstruction/ obstructive syndrome/intestinal obstruction at the initial diagnosis receives clear (surgical) therapy to resolve symptoms, the subject may be enrolled;
* Evidence on intraperitoneal pneumatosis that can not be explained by puncture or recent surgery;
* Previous or current presence of metastasis to central nervous system;
* Previous or present history of pulmonary fibrosis, organising pneumonia (e.g., obliterative bronchiolitis), interstitial pneumonia, pneumoconiosis, drug related pneumonitis, idiopathic pneumonia, or allowable previous radiation pneumonitis in the radiation area (fibrosis) for subjects with evidence on active pneumonia or serious pulmonary function impairment on thoracic computed tomography (CT) in screening period that may interfere with the detection and treatment of suspected drug related pulmonary toxicity; active tuberculosis;
* Any active autoimmune disease or history of autoimmune disease and expected recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects that can be controlled with hormone replacement therapy only can be enrolled]); subjects with skin diseases that does no need systemic treatment, for example, leukoderma, psoriasis, alopecia, those with controlled type I diabetes by insulin or those with asthma that has been completely resolved in childhood and with no need of any intervention can be enrolled; while subjects with asthma who need bronchodilator for medical intervention can not be enrolled;
* Current use of immunosuppressive medication, or systemic corticosteroid therapy to achieve the objective of immunosuppression (Prednisone at the dose of >10mg/day or equivalent), and continuous use within two weeks prior signing informed consent form;
* Use of strong CYP3A4/CYP2C19 inducers, including rifampicin (and its analogues) and St. Jonhn's Wort, or strong CYP3A4/CYP2C19 inhibitors within two weeks prior to the signature of informed consent form;
* Known history of serious allergy to any monoclonal antibody or targeted anti-angiogenic drug;
* Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia or complications of severe pneumonia; oral or intravenous therapeutic antibiotics within two weeks prior to the start of study treatment (for example, subjects who are given with preventive antibiotics for prevention of urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible for participation in the study);
* Congenital or acquired immunodeficiency (e.g., HIV infection);
* Combined hepatitis B and hepatitis C co-infection;
* Previous treatment with other PD-1 antibody or other immunotherapy against PD-1/PD-L1, or previous use of other small molecules of anti-angiogenesis TKI drugs, such as pazopanib, sorafenib;
* Palliative radiotherapy for non-target lesions to control symptoms is allowed, but it must be completed at least 2 weeks prior to the start of study treatment, and the adverse event induced by radiotherapy must have resolved/improved to ≤CTCAE Grade 1;
* Treatment of other investigational product(s) within 28 days prior to the start of study treatment;
* Other factors that may affect the study results or lead to forced termination of the study early as judged by investigators, such as alcoholism, drug abuse, other serious diseases (including mental disorders) requiring concomitant therapy, with serious laboratory examination abnormality, with family or social factors, that may affect subject's safety.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months
  CR+PR according to RECIST 1.1
Progression-free Survival, PFS | 6 months
  Progression-free survival is defined as time from randomisation to the first occurrence of progression of disease or death from any cause within 63 days of last response assessment or randomisation.

SECONDARY OUTCOMES:
Overall Survival, OS | 12 months
  Overall survival is was defined as time from randomisation to the first occurrence of death from any cause within 63 days of last response assessment or randomisation. randomisation to the first occurrence of progression of disease orrandomisation.
Duration of response, DOR | 6 months
  Duration of response is defined as from the time of occurence of best overall response to progression or death for the proportion of patients achieving an overall response.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Ph.D. and M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University Shougang Hospital
Locations (1):
- Lu Xie, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie L, Xu J, Sun X, Tang X, Yan T, Yang R, Guo W. Apatinib for Advanced Osteosarcoma after Failure of Standard Multimodal Therapy: An Open Label Phase II Clinical Trial. Oncologist. 2019 Jul;24(7):e542-e550. doi: 10.1634/theoncologist.2018-0542. Epub 2018 Dec 17. PMID 30559126
- [Background] Xie L, Guo W, Wang Y, Yan T, Ji T, Xu J. Apatinib for advanced sarcoma: results from multiple institutions' off-label use in China. BMC Cancer. 2018 Apr 6;18(1):396. doi: 10.1186/s12885-018-4303-z. PMID 29625604